CLINICAL TRIAL: NCT01960907
Title: Clinical Trials for Elderly Patients With Multiple Disease
Acronym: CHROMED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Restech Srl (Industry)
Collaborators: University of Liverpool (Other); Uppsala University (Other); University of Lincoln (Other); University of Tallin (Unknown); University of Barcelona (Other); Hospital of Sezana (Unknown); University Hospital of North Norway (Other); Tesan spa (Unknown)
Responsible Party: Principal Investigator, Pasquale Pio Pompilio, PhD, Restech Srl
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHROMEDB
Record Dates: First submitted 2013-10-09; First posted 2013-10-11 (Estimated); Results first posted 2016-09-30 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Congestive Heart Failure (CHF); Sleep Disordered Breathing (SDB)
Keywords: COPD; CHF; SDB
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Heart Failure; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Observational (No Intervention): Subjects in the observational arm will receive monthly interviews for collecting informations about their status and level of utilization of healthcare resources.
  They will follow their usual care path as provided by their local NHS
- Interventional (Experimental): Patients will receive a system form monitoring their health status.
  The system is composed by:
  * a touch-screen pc for the administration of daily questionnaires
  * RESMONPRO DIARY for the measurement of lung mechanical impedance and breathing pattern
  * a Medic4all Wrist Clinic for the assessment of heart rate, blood pressure, saturation, 1 lead ECG, body temperature.
  Subjects will receive medical treatment following the activation of alarms by the monitoring devices.
  Monthly phone interviews will be performed to collect data about their level of utilization of the health care system.
  Interventions: Device: CHROMED monitoring system

INTERVENTIONS:
Device: CHROMED monitoring system — Optimization of patient's treatment according to the data collected by the home monitoring devices
  Arms: Interventional

SUMMARY:
The CHROMED project focuses its investigation on the applicability of an integrated solution for a pathological condition which: a) is very prevalent in ageing patients and b) severely impairs quality of life: COPD with other typical comorbidities such as congestive heart failure and sleep disordered breathing. A specific ICT platform in combination with a set of innovative devices will be used to collect and process useful clinical data at the patient's home and used to optimize their medical treatment. To evaluate the impact of this solution, an international multi-centric randomized control trial will be implemented in five European regions: United Kingdom, Sweden, Estonia, Spain and Slovenia, representing different social and organizational contexts in Europe.

ELIGIBILITY:
Inclusion Criteria:

* COPD GOLD grade II or higher with a prior history of exacerbations and/or an hospitalization for COPD in the previous year with one or more documented non-pulmonary chronic conditions such as:
* CHF due to left ventricular systolic dysfunction (LVSD) confirmed on echocardiography
* SDB identified by respiratory sleeping studies or polysomnography
* current or prior smoking history of >= 10 pack/years
* subjects capable of providing signed written informed consent
* subjects capable of perform study procedures and use the RESMONPRO at home
* subjects with reliable mobile phone coverage at home

Exclusion Criteria:

* Any disease that, in the opinion of the investigator, put the subject at risk
* subjects with significant vision disturbance and mental diseases
* subjects with a planned prolonged absence from home

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 312 (Actual)
Dates: Start 2013-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Calverley, Phd, MD, Principal Investigator — University of Liverpool
Locations (6):
- Institute of Clinical Medicine, Tallinn, Estonia
- Bolnisnica Sežana Zavod, Sežana, Slovenia
- Hospital clinic, Barcelona, Spain
- Uppsala University Hospital, Uppsala, Sweden
- United Kingdom (2):
  - Lincolnshire Community Health Service, Lincoln
  - Aintree University Hospital, Liverpool

REFERENCES:
- [Background] Brouwer AF, Visser CA, Duiverman EJ, Roorda RJ, Brand PL. Is home spirometry useful in diagnosing asthma in children with nonspecific respiratory symptoms? Pediatr Pulmonol. 2010 Apr;45(4):326-32. doi: 10.1002/ppul.21183. PMID 20196110
- [Background] Dellaca RL, Santus P, Aliverti A, Stevenson N, Centanni S, Macklem PT, Pedotti A, Calverley PM. Detection of expiratory flow limitation in COPD using the forced oscillation technique. Eur Respir J. 2004 Feb;23(2):232-40. doi: 10.1183/09031936.04.00046804. PMID 14979497
- [Background] Dellaca RL, Pompilio PP, Walker PP, Duffy N, Pedotti A, Calverley PM. Effect of bronchodilation on expiratory flow limitation and resting lung mechanics in COPD. Eur Respir J. 2009 Jun;33(6):1329-37. doi: 10.1183/09031936.00139608. Epub 2009 Jan 22. PMID 19164347
- [Background] Dellaca R, Montserrat JM, Govoni L, Pedotti A, Navajas D, Farre R. Telemetric CPAP titration at home in patients with sleep apnea-hypopnea syndrome. Sleep Med. 2011 Feb;12(2):153-7. doi: 10.1016/j.sleep.2010.07.014. Epub 2011 Jan 17. PMID 21247800
- [Background] Wilkinson TM, Donaldson GC, Hurst JR, Seemungal TA, Wedzicha JA. Early therapy improves outcomes of exacerbations of chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2004 Jun 15;169(12):1298-303. doi: 10.1164/rccm.200310-1443OC. Epub 2004 Feb 27. PMID 14990395
- [Background] McKinstry B, Pinnock H, Sheikh A. Telemedicine for management of patients with COPD? Lancet. 2009 Aug 29;374(9691):672-3. doi: 10.1016/S0140-6736(09)61542-7. No abstract available. PMID 19716948
- [Background] Feary JR, Rodrigues LC, Smith CJ, Hubbard RB, Gibson JE. Prevalence of major comorbidities in subjects with COPD and incidence of myocardial infarction and stroke: a comprehensive analysis using data from primary care. Thorax. 2010 Nov;65(11):956-62. doi: 10.1136/thx.2009.128082. Epub 2010 Sep 25. PMID 20871122
- [Background] Vinson JM, Rich MW, Sperry JC, Shah AS, McNamara T. Early readmission of elderly patients with congestive heart failure. J Am Geriatr Soc. 1990 Dec;38(12):1290-5. doi: 10.1111/j.1532-5415.1990.tb03450.x. PMID 2254567
- [Background] MacDonald M, Fang J, Pittman SD, White DP, Malhotra A. The current prevalence of sleep disordered breathing in congestive heart failure patients treated with beta-blockers. J Clin Sleep Med. 2008 Feb 15;4(1):38-42. PMID 18350960
- [Background] Polisena J, Tran K, Cimon K, Hutton B, McGill S, Palmer K, Scott RE. Home telehealth for chronic obstructive pulmonary disease: a systematic review and meta-analysis. J Telemed Telecare. 2010;16(3):120-7. doi: 10.1258/jtt.2009.090812. Epub 2010 Mar 2. PMID 20197355
- [Background] Rutten FH, Cramer MJ, Lammers JW, Grobbee DE, Hoes AW. Heart failure and chronic obstructive pulmonary disease: An ignored combination? Eur J Heart Fail. 2006 Nov;8(7):706-11. doi: 10.1016/j.ejheart.2006.01.010. Epub 2006 Mar 13. PMID 16531114
- [Background] Calverley P, Pauwels Dagger R, Lofdahl CG, Svensson K, Higenbottam T, Carlsson LG, Stahl E. Relationship between respiratory symptoms and medical treatment in exacerbations of COPD. Eur Respir J. 2005 Sep;26(3):406-13. doi: 10.1183/09031936.05.00143404. PMID 16135720
- [Background] Spencer S, Calverley PM, Burge PS, Jones PW. Impact of preventing exacerbations on deterioration of health status in COPD. Eur Respir J. 2004 May;23(5):698-702. doi: 10.1183/09031936.04.00121404. PMID 15176682
- [Background] McNicholas WT. Chronic obstructive pulmonary disease and obstructive sleep apnea: overlaps in pathophysiology, systemic inflammation, and cardiovascular disease. Am J Respir Crit Care Med. 2009 Oct 15;180(8):692-700. doi: 10.1164/rccm.200903-0347PP. Epub 2009 Jul 23. PMID 19628778
- [Background] Johnson MK, Birch M, Carter R, Kinsella J, Stevenson RD. Measurement of physiological recovery from exacerbation of chronic obstructive pulmonary disease using within-breath forced oscillometry. Thorax. 2007 Apr;62(4):299-306. doi: 10.1136/thx.2006.061044. Epub 2006 Nov 14. PMID 17105778
- [Derived] Middlemass JB, Vos J, Siriwardena AN. Perceptions on use of home telemonitoring in patients with long term conditions - concordance with the Health Information Technology Acceptance Model: a qualitative collective case study. BMC Med Inform Decis Mak. 2017 Jun 26;17(1):89. doi: 10.1186/s12911-017-0486-5. PMID 28651588

RESULTS

PARTICIPANT FLOW:
Groups:
- Observational: Subjects in the observational arm received monthly interviews for collecting informations about their status and level of utilization of healthcare resources.
  They followed their usual care path as provided by their local NHS.
- Interventional: Patients received a system for monitoring their health status.
  The system is composed by:
  * a touch-screen pc for the administration of daily questionnaires
  * RESMON PRO DIARY for the measurement of lung mechanical impedance and breathing pattern
  * a Medic4all Wrist Clinic for the assessment of heart rate, blood pressure, saturation, 1 lead ECG, body temperature.
  Subjects received medical treatment following the activation of alarms by the monitoring devices.
  Monthly phone interviews were performed to collect data bout their status and level of utilization of healthcare resources.
Period: Overall Study
Arm/Group | Observational | Interventional
Started | 158 | 154
Completed | 122 | 109
Not Completed | 36 | 45
Not completed — Death | 4 | 3
Not completed — Withdrawal by Subject | 32 | 42

BASELINE CHARACTERISTICS:
Groups:
- Interventional: Patients received a system for monitoring their health status.
  The system is composed by:
  * a touch-screen pc for the administration of daily questionnaires
  * RESMON PRO DIARY for the measurement of lung mechanical impedance and breathing pattern
  * a Medic4all Wrist Clinic for the assessment of heart rate, blood pressure, saturation, 1 lead ECG, body temperature.
  Subjects received additional medical treatment following the activation of alarms by the monitoring devices.
  Monthly phone interviews were performed to collect data bout their status and level of utilization of healthcare resources.
- Total: Total of all reporting groups
Arm/Group | Observational | Interventional | Total
Number analyzed (Participants) | 158 | 154 | 312
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 71 [65.3 to 76] | 71 [66 to 75.8] | 71 [66 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 53 | 106
  Male | 105 | 101 | 206
Region of Enrollment [Number; unit: participants]
  Sweden | 32 | 31 | 63
  United Kingdom | 41 | 34 | 75
  Slovenia | 16 | 17 | 33
  Estonia | 39 | 41 | 80
  Spain | 30 | 31 | 61
FEV1 postBD [Median (Inter-Quartile Range); unit: L] — Spirometrically measured Forced Exhaled Volume in 1 second (FEV1), measured after a maximal dose of a bronchodilator drug
  L | 1.3 [0.9 to 1.8] | 1.3 [1.0 to 1.6] | 1.3 [1.0 to 1.7]
FEV1 postBD %pred [Median (Inter-Quartile Range); unit: %predicted] — Forced Exhaled Volume in 1 second (FEV1) measured after the administration of a maximal dose of bronchodilator expressed as percentage of predicted value.
  %predicted | 50.4 [38 to 63.9] | 49.4 [37.1 to 59.2] | 49.8 [37.2 to 62.1]
FVC postBD [Median (Inter-Quartile Range); unit: L] — Forced Vital Capacity (FVC) after brochodilation: maximum volume of air exhaled during a full forced exhalation from the maximum to the minimum lung volume achievable by the subject measured after the administration of a maximal dose of a bronchodilator drug.
  L | 2.5 [2.1 to 3.1] | 2.6 [2.0 to 3.1] | 2.5 [2.0 to 3.1]
FVC postBD %pred [Median (Inter-Quartile Range); unit: %predicted] — Forced Vital Capacity measured after bronchodilation expressed as percentage of its predicted value.
  %predicted | 75.8 [63.0 to 89.7] | 73.8 [61.8 to 88.0] | 75.0 [62.2 to 89.0]
FEV1/FVC postBD [Median (Inter-Quartile Range); unit: ratio] — Ratio between Forced Exhaled Volume in 1 second (FEV1) and the Forced Vital capacity (FVC)
  ratio | 0.5 [0.4 to 0.6] | 0.5 [0.4 to 0.6] | 0.5 [0.4 to 0.6]
Patients with two or more COPD exacerbation in the previous year [Number; unit: participants] | 99 | 91 | 190
Patients with one or more hospitalization in the previous year [Number; unit: participants] | 65 | 64 | 129

OUTCOME MEASURES:

1. Primary Outcome: Time to First Hospitalization
Description: It represents the number of days, since the enrolment into the study, to the first hospitalization
Time Frame: From enrolment up to 9 months
Population: An intention to treat analysis has been applied for the primary outcomes of the trial and all the randomized patients have been retained for the analysis.
Measure: Mean (Inter-Quartile Range); unit: days
Arm/Group | Observational | Interventional
Number analyzed (Participants) | 158 | 154
days | 255 [240 to 270] | 224 [209 to 240]
Statistical Analysis 1: Comparison: Observational vs Interventional; Test type: Superiority or Other; p = 0.342, Log Rank

2. Primary Outcome: Final Utility Index of EQ-5D Questionnaire
Description: The quality of life of patients as quantified by the final utility index of the EQ-5D questionnaire. The utility index ranges from -0.074 to 1 with 1 being the highest possible quality of life.
Time Frame: 9 months
Population: An intention to treat analysis has been applied for the primary outcomes of the trial. Multiple Imputation (MI) was used to assign values were data were missing. However for a limited number of patient, due to the fact that all data were missing, we couldn't apply any imputation method and therefore they have been excluded.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Observational | Interventional
Number analyzed (Participants) | 153 | 150
units on a scale | 0.640 (0.248) | 0.637 (0.225)
Statistical Analysis 1: Comparison: Observational vs Interventional; Test type: Superiority or Other; p = 0.915, t-test, 2 sided

3. Post Hoc Outcome: Difference of Hospitalization Rate
Description: Difference between the hospitalization rate during the study and the previous year. For each patient, hospitalization rate was defined as the number of hospital admissions during a period divided by the length (in days) of the period. Number of hospitalizations was collected by the hospital clinical records.
Time Frame: Baseline and 9 months
Measure: Median (Inter-Quartile Range); unit: hospitalizations/year/patient
Groups:
- Monitored, Previously Hopitalized for COPD Exacerbation: Patients in the monitored group that were hospitalized the year before the study for a COPD exacerbation
- Observational, Previously Hopitalized for COPD Exacerb.: Patients in the observational group that were hospitalized the year before the study for a COPD exacerbation
Arm/Group | Monitored, Previously Hopitalized for COPD Exacerbation | Observational, Previously Hopitalized for COPD Exacerb.
Number analyzed (Participants) | 64 | 65
hospitalizations/year/patient | -1 [-1 to -0.15] | -1 [-1 to 1.04]
Statistical Analysis 1: Comparison: Monitored, Previously Hopitalized for COPD Exacerbation vs Observational, Previously Hopitalized for COPD Exacerb; Test type: Superiority or Other; p = 0.038, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Observational | Interventional
Serious Adverse Events (participants affected / at risk) | 0/158 | 0/154
Other Adverse Events (participants affected / at risk) | 0/158 | 0/154

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No